CLINICAL TRIAL: NCT04063475
Title: Cyanoacrylate Tissue Adhesive Assisted Soft Tissue Stabilization: a Novel Technique for Free Gingival Graft Fixation (Case Series Study)
Brief Title: Cyanoacrylate With Sutures for Fixation of Free Gingival Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, haytham mohamed ahmed ibrahim, student, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: cyanoacrylate in FGG
Record Dates: First submitted 2019-06-16; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-06

CONDITIONS: Soft Tissue Atrophy
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Intervention Model Description: Cyanoacrylate beside sutures for Fixation of FGG
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cyanoacrylate beside sutures for FGG fixation (Experimental): butyl cyanoacrylate
  Interventions: Drug: cyanoacrylate tissue adhesive beside sutures

INTERVENTIONS:
Drug: cyanoacrylate tissue adhesive beside sutures — using cyanoacrylate tissue adhesive for FGG fixation
  Other Names: tissue adhesive

SUMMARY:
fixation of FGG with sutures alone is not sufficient,we use cyanoacrylate beside sutures for fixation

DETAILED DESCRIPTION:
Inadequate zone of attached mucosa around implants, gingival recession, inadequate ridge width or height despite there is enouph bone for implant placement are problems that face periodontists and can be treated by soft tissue graft Studies have demonstrated the importance of the tissues stability for the first hours when support is provided by underlying osseous or dental structures.

Movement of the graft during mastication and phonation will disturb healing procedures. Most of the clinicians prefer a protective device during the healing phase.

Transitional dentures are not stable themselves, and hence are not suitable for stabilizing.

Circummandibular wiring and impact posts are seemingly very aggressive for patients and need extra clinical practices, skills, and equipment.

Studies proved that the maximum tissue shrinkage (approximately 20%-40%) occurs during the first 3 months post operation and will proceed until 12 postsurgical months with a persistent, significantly lower rate.

In this study we give more stabilization for free gingival grafts by using cyanoacrylate tissue adhesive beside sutures Its autogenous character, maintenance of keratinization, predictability, ease of technique tlead CTG to be accepted as the golden standard to increase attached gingival dimensions Cyanoacrylate is a simple, inexpensive haemostatic and biocompatible material It is used as tissue adhesives in paediatric surgery general surgery and also dentistry.

it has been applied intraorally with different purposes such as periodontal dressing,for sealing sinus membrane perforations for stabilizing bone fragments during fracture fixation, and in closing peripheral nerve anastomosis it seems promising in the intraoral field due to their strong sealing, bacteriostatic, and hemostatic properties. Multiple studies examined the use of cyanoacrylate glues as an alternative to suturing intraoral and extraoral wounds concluding that cyanoacrylates are faster, more reliable ,and less painful and cause better hemostasis .

ELIGIBILITY:
Inclusion Criteria:

* Patients with hopeless teeth that need extraction
* Age: between 20 and 60 years
* Both sexes.
* Subjects willing to sign an informed consent form ,participate in the study and return for follow-up visits

Exclusion Criteria:

* • Patients with coagulation disorders (Hemophilia a/b, von Willebrand disease, liver disease, anticoagulative therapy),

  * patients on corticosteroids,
  * patients with uncontrolled diabetes mellitus
  * smokers
  * Pregnant or lactating mother.
  * Known systemic diseases and/ or drug therapy which may interfere with wound healing or contraindicate periodontal therapy
  * Allergy to cyanoacrylate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-16 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
graft shrinkage in millimeter | 2 weeks,month,3months
  graft area ,thickness in millimeter

SECONDARY OUTCOMES:
success percentage | 3 months
  % percentage (success of Free Gingival Graft Fixation)

IPD SHARING:
Plan to Share IPD: No